CLINICAL TRIAL: NCT04188639
Title: Emicizumab in Patients With Acquired Hemophilia A: Multicenter, Single-arm, Open-label Clinical Trial
Brief Title: Emicizumab in Acquired Hemophilia A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Hoffmann-La Roche (Industry); Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHA-EMI (MO41153)
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Hemophilia A, Acquired
Keywords: acquired Hemophilia A; Factor VIII activity; Emicizumab
MeSH Terms: conditions — Factor 8 deficiency, acquired | interventions — emicizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with emicizumab (Experimental)
  Interventions: Drug: Emicizumab Injection

INTERVENTIONS:
Drug: Emicizumab Injection — All eligible patients with AHA will receive the same study medication consisting of once weekly subcutaneous emicizumab. For each subject, the maximal duration of the study will be 24 weeks including 12 weeks treatment with emicizumab and 12 weeks follow-up with Immunosuppressive therapy (IST) at the investigators discretion.
  Other Names: Hemlibra (R)

SUMMARY:
This study is an international, multicenter, open-label, single arm, prospective clinical trial and will evaluate the efficacy of prophylactic emicizumab administered on a scheduled basis to prevent bleeds in patients with acquired hemophilia A (AHA).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AHA based on a reduced FVIII activity (<50 %) and positive FVIII inhibitor (>0.6 BU/ml) (local laboratory) at time of diagnosis
* Signed informed consent form by the participant or a Person who is legally authorized to sign on behalf of the participant before any study specific tests or procedures are done
* Male or female patients aged 18 years or older at the time of informed consent
* Ability to understand and follow study-related instructions
* Current bleeds due to AHA at the time of screening

Exclusion Criteria:

* Congenital hemophilia A
* Partial or complete remission of AHA (defined as FVIII activity ≥ 50 % and no bleeding and no hemostatic therapy) at the time of screening
* Treatment with aPCC within the last 48 h before first study treatment or planned treatment with aPCC during the course of the study
* Treatment of AHA within the days before study enrollment with more than 100 mg prednisolone (or equivalent) per day or prednisolone for more than 2 days or with other immunosuppressive drugs (e.g. rituximab, cyclophosphamide). IST for other concomitant disorders (e.g. autoimmune disorders) is not an exclusion criterion and can be continued at the investigator's discrétion
* Therapy (current or planned during the emicizumab treatment period) with immunosuppressive or immune modulating drugs that were not already given on a regular basis before first diagnosis of AHA
* Positive lupus anticoagulant at the time of screening
* Severe uncontrolled infection at the time of screening
* Signs of active disseminated intravascular coagulation at the time of screening
* Current treatment for thromboembolic disease or signs of current thromboembolic disease at time of screening
* Patients who are at high risk for TMA (e.g., have a previous medical or family history of TMA), in the investigator's judgment
* Known severe congenital or acquired thrombophilia
* Life expectancy <3 months at the time of screening
* Other conditions that substantially increase risk of bleeding or thrombosis by the discretion of the investigator
* Contraindications according to the local SmPC of emicizumab (see 16.1 Appendix I)
* Current treatment with emicizumab at time of screening
* History of clinically significant hypersensitivity associated with monoclonal antibody therapies or components of the emicizumab injection by the discretion of the investigator
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study, may pose additional risk, or would, in the opinion of the local investigator, preclude the patient's safe participation in and completion of the study
* Addiction or other diseases that preclude the patient from appropriately assessing the nature and scope as well as possible consequences of the clinical study by the discretion of the investigator
* Pregnant or breast-feeding women
* Women of childbearing potential unless women who meet the following criteria:

  1. Post-menopausal (12 months natural amenorrhea or 6 months amenorrhea with serum FSH > 40 U/mL)
  2. Postoperatively (six weeks after bilateral ovariectomy with or without hysterectomy)
  3. Regular and correct use of a contraceptive method with error rate <1% per year such as implants, depot injections, oral contraceptives or intrauterine devices
  4. Sexual abstinence
  5. Vasectomy of the partner
* Men of sexual activity with women of childbearing potential who are not willing to use an effective barrier method of contraception during and up to 3 months after the end of therapy
* Subject is in custody by order of an authority or a court of law
* Receipt of an investigational drug concurrently or within 5 half-lives before administration of the study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
The number of clinically significant bleeds per patient-week until death or week 12 after starting emicizumab treatment, whatever occurs first | 12 weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events, thromboembolic events, thrombotic microangiopathy in the 12 weeks after starting emicizumab | 12 weeks
Incidence of mortality and cause of death in the 24 weeks after starting emicizumab treatment | 24 weeks
Days of treatment with and total dose of bypassing agents (recombinant factor VIIa, activated prothrombin complex concentrate) or recombinant porcine factor VIII (susoctocag alfa) or other factor VIII concentrates | 24 weeks
Days in hospital during 12 weeks of emicizumab treatment | 12 weeks
Number of patients achieving partial remission in the 24 weeks after starting emicizumab treatment | 24 weeks
Bleeding-free survival in the 12 weeks after starting emicizumab treatment | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Tiede, Prof. Dr., Study Director — Hannover Medical School
Locations (16):
- Austria (3):
  - Medizinische Universität Wien, Hämatologie/Hämostaseologie, Wien, Lower Austria
  - Medizinische Universitätsklinik Graz, Graz, Styria
  - Landeskrankenhaus Salzburg, Universitätsklinikum der PMU, Innere Med. III, Salzburg
- Germany (13):
  - LMU Klinikum, Hämophiliezentrum Erwachsene/Transfusionsmedizin, München, Bavaria
  - Universitätsklinikum Regensburg, Innere Med. III - Studienzentrale, Regensburg, Bavaria
  - Universitätsklinikum Frankfurt, Hämostaseologie/Hämophiliezentrum, Frankfurt am Main, Hesse
  - Universitätsklinikum Gießen und Marburg, Giessen, Hesse
  - Medizinische Hochschule Hannover, Hämatologie/Hämostaseologie, Hanover, Lower Saxony
  - Universitätsklinikum Bonn, Hämatologie/Transfusionsmedizin/Hämophilie, Bonn, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Institut für Klinische Hämostaseologie und Transfusionsmedizin, Homburg / Saar, Saarland
  - Universitätsklinikum Dresden, Med. Poliklinik I, Dresden, Saxony
  - Universitätsklinikum Leipzig, Medizinische Klinik und Poliklinik I, Bereich Hämostaseologie, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein, Klinische Chemie/Gerinnungszentrum, Kiel, Schleswig-Holstein
  - Vivantes Klinikum im Friedrichshain, Angiologie/Hämostaseologie, Friedrichshain, State of Berlin
  - Universitätsklinikum Jena, Klinik für Innere Medizin II, Jena, Thuringia
  - Universitätsklinikum Hamburg-Eppendorf, Med. Klinik II/Gerinnungsambulanz, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schimansky IM, Dobbelstein C, Klamroth R, Hart C, Sachs UJ, Greil R, Knobl P, Oldenburg J, Miesbach W, Pfrepper C, Trautmann-Grill K, Mohnle P, Holstein K, Eichler H, Werwitzke S, Tiede A. Sustained survival benefit of emicizumab and postponed immunosuppression in acquired hemophilia A. Blood Adv. 2025 Nov 25;9(22):5853-5860. doi: 10.1182/bloodadvances.2025017144. PMID 40795229
- [Derived] Tiede A, Hart C, Knobl P, Greil R, Oldenburg J, Sachs UJ, Miesbach W, Pfrepper C, Trautmann-Grill K, Holstein K, Pilch J, Mohnle P, Schindler C, Weigt C, Schipp D, May M, Dobbelstein C, Pelzer FJ, Werwitzke S, Klamroth R. Emicizumab prophylaxis in patients with acquired haemophilia A (GTH-AHA-EMI): an open-label, single-arm, multicentre, phase 2 study. Lancet Haematol. 2023 Nov;10(11):e913-e921. doi: 10.1016/S2352-3026(23)00280-6. Epub 2023 Oct 16. PMID 37858328